CLINICAL TRIAL: NCT00355628
Title: Phase II Clinical Study of KW-2246 in Patients With Cancer Pain - Maintenance Switch Study in Oral Morphine or Oral Oxycodone-treated Patients
Brief Title: Clinical Study of KW-2246 in Patients With Cancer Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2246-0401
Record Dates: First submitted 2006-07-21; First posted 2006-07-24 (Estimated); Last update posted 2012-08-31 (Estimated); Status verified 2012-08

CONDITIONS: Pain; Cancer
Keywords: Pain; Cancer; Neoplasm; Continual Reassessment Method; Pain Associated with Cancer/Neoplasms
MeSH Terms: conditions — Pain; Neoplasms | interventions — Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): KW-2246 (fentanyl citrate)
  Interventions: Drug: KW-2246 (fentanyl citrate)

INTERVENTIONS:
Drug: KW-2246 (fentanyl citrate) — KW-2246
  Other Names: Fentanyl citrate

SUMMARY:
This study is a Phase II open-label study to investigate the recommended conversion ratio (oral morphine dose to KW-2246) when switching oral morphine or oxycodone to KW-2246 in cancer patients.

DETAILED DESCRIPTION:
This study is a Phase II open-label study to investigate, using the continual reassessment method procedure by pain intensity and safety as indicators, the recommended conversion ratio (oral morphine dose to KW-2246) when switching oral morphine or oxycodone to KW-2246 in cancer patients who have been maintained on oral morphine or oral oxycodone for pain and to evaluate the safety and efficacy of KW-2246.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent to participate in the study.
2. Be able to be hospitalized.
3. Between the ages of 20 and 80 years (inclusive) at the time of giving written informed consent.
4. Have regularly received oral morphine or oral oxycodone at an oral morphine equivalent dose of 20 to 120 mg/day for at least 2 days before study entry, AND not have required any rescue dose between regular doses.
5. Not have experienced intolerable toxicity for 2 days before study entry.
6. Have cancer that is in stable condition at study entry and expected to remain stable during the KW-2246 treatment period.
7. Have a life expectancy of at least 1 month after the start of KW-2246 administration.
8. Considered to be able to keep the patient diary.

Exclusion Criteria:

1. Serious respiratory dysfunction.
2. Asthma.
3. Serious bradyarrhythmia.
4. Serious hepatic or renal dysfunction.
5. Susceptibility to respiratory depression due to such conditions as increased intracranial pressure, head injury and brain tumor.
6. History of convulsive seizures (except a single episode of infantile febrile convulsions).
7. Current or past history of drug dependence or narcotic abuse.
8. Dry mouth that affects oral intake.
9. Use of opioid analgesics other than oral morphine or oxycodone within 7 days prior to study entry.
10. Use of narcotic antagonists within 7 days prior to study entry.
11. Interventions that may affect pain evaluation, such as surgery, radiation to the pain site (including those sites that influence pain) and nerve block, within 7 days prior to study entry or scheduled to be given during the study.
12. Patients with a history of serious adverse reactions to the combination of opioid analgesics and other drugs/substances who are currently receiving or expected to receive those drugs/substances combined to opioid analgesics.
13. History of hypersensitivity to fentanyl.
14. Pregnant or lactating women, possibly pregnant women or women who are planning to become pregnant.
15. Participation in any other clinical trial within 28 days prior to the start of KW-2246 treatment.
16. Prior exposure to KW-2246.
17. Patients whom an investigator judge unsuitable for enrollment.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2006-07; Primary Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability | At every visit
Pain Intensity as Rated on a Categorical Scale | At specified visits

SECONDARY OUTCOMES:
Pain Intensity as Rated on a Visual Analog Scale (VAS) | At specified visits
Number of Rescue Doses per Day | At every visit
Regular Dose Level of KW-2246 | At every visit

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Kyowa Kirin Co., Ltd.
Locations (1):
- Nagoya Medical Center, Nagoya, Japan